CLINICAL TRIAL: NCT06237816
Title: CTNow: A Clinical Trials Education Program for Rural Cancer Patients and Oncology Providers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Okado-2023-2
Record Dates: First submitted 2023-12-07; First posted 2024-02-02 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Intervention (Experimental): A multimedia educational series is designed to provide patient education on cancer clinical trials.
  The following topics are addressed:
  * What is a clinical trial?
  * Types of clinical trials.
  * Phases of clinical trials.
  * Benefits and drawbacks.
  * Costs.
  * FAQs. This section covers common myths and clarifies these myths using a Q&A format.
  * How to join a clinical trial. Information about eligibility and informed consent.
  * Clinical trial stories. Testimonies from oncology providers and patients. Each module is approximately 2-5 minutes, and they can be reviewed in the order/schedule preferred by the patient.
  The overall program is 30 minutes to view including the videos. The tablet provided to patients provides additional benefits for participation.
  Interventions: Other: Patient Education Intervention
- Provider Education Intervention (Experimental): The provider education intervention will consist of 3 provider informational sessions conducted individually. These individual provider sessions will be conducted by teleconference by the research team and scheduled according to provider's availability.
  Provider workshops are designed to provide both a background on clinical trial infrastructure in Hawaii and resources for additional information. The content of these sessions includes:
  * An overview of clinical trials infrastructure in Hawaii.
  * Available trials in Hawaii. At each informational session, the research team will review available trials and any new/upcoming trials with the provider.
  * An overview of how to get involved in clinical trials. As experience and background re: clinical trials may vary across providers, the content of these informational sessions will be tailored to each provider. Following the initial session, 2 additional meetings will be scheduled in 4-6 months as follow-up sessions.
  Interventions: Other: Provider Education Intervention

INTERVENTIONS:
Other: Patient Education Intervention — Multimedia Educational Videos
  Arms: Patient Education Intervention
Other: Provider Education Intervention — Provider workshops via zoom
  Arms: Provider Education Intervention

SUMMARY:
The overall goal of the project is to pilot test CTNow, a multilevel intervention designed to facilitate access and referrals to cancer clinical trials in rural areas through patient and provider education and teleconference resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with any cancer.
* Patients who have received treatment, are receiving cancer treatment at the time of enrollment, or estimated to start treatment within 90 days.
* Patients must be ≥ 18 years of age. Patients must be able to read, write, and speak English. Study materials and telephone calls are only available in English.

Patients must be residents of Hawaii, Kauai, or Maui counties.

Exclusion Criteria:

* Patients must not have previously participated in a cancer clinical trial. Those who have participated in a cancer clinical trial are not eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in patients' awareness and knowledge of clinical trials | 18 months
  Participants will complete a 12-item awareness and knowledge of clinical trials questionnaire at baseline and post-intervention. Items are reported on a Likert-type scale , with higher scores indicating greater knowledge. A paired t-test will be used to evaluate whether there is a statistically significant difference in pre- and post-intervention scores on patients' knowledge of clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Izumi Okado, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- Univesity of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No